CLINICAL TRIAL: NCT02011685
Title: Practice-Based Trial of Home BP Telemonitoring Among Minority Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-00281; U54NS081765-5162 (Other: National Institute of Neurological Disorders and Stroke (NINDS)); U54NS081765 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Stroke; Hypertension
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home BP Telemonitoring (HBPTM) (Active Comparator): Participants will take home BP readings 3 days per week (morning and evening) for one week out of each month during the 12-month intervention.
  Interventions: Behavioral: Home BP Telemonitoring (HBPTM)
- HBPTM + Nurse Case Management (NCM) (Experimental): Participants will complete the same Home BP Telemonitoring protocol and will also complete 20 counseling phone calls with a nurse case manager during the 12-month intervention.
  Interventions: Behavioral: Home BP Telemonitoring (HBPTM); Behavioral: Nurse Case Management (NCM)

INTERVENTIONS:
Behavioral: Home BP Telemonitoring (HBPTM) — Participants will take home BP readings 3 days per week (morning and evening), one week out of every month for 12 months. BP readings will be transmitted wirelessly to a secure server. Patients' physicians will receive home BP reports via secure email before every scheduled appointment for the duration of the study to facilitate necessary treatment intensification and medication adjustments.
Behavioral: Nurse Case Management (NCM) — Participants will complete 20 counseling phone calls with a nurse case manager (NCM) during the 12-month intervention: weekly calls for Months 1-2; biweekly calls for Months 3-4; and monthly calls for Months 5-12. The NCMs will provide self-management education, medication and appointment reminders, and will facilitate patient-provider communication. They will counsel patients on specific self-management behaviors using problem solving and motivational interviewing techniques. Target behaviors will include dietary changes, physical activity, weight loss, medication adherence, and smoking cessation. NCMs will also review patients' clinical information and provide feedback about abnormal lab results, and will communicate with the patient's physician as needed (e.g., regarding barriers).
  Arms: HBPTM + Nurse Case Management (NCM)

SUMMARY:
This study will assess the comparative effectiveness, cost-effectiveness and sustainability of two telemonitoring interventions in reducing blood pressure and recurrent stroke among 450 high-risk Black and Hispanic stroke patients. The primary hypothesis is that home blood pressure telemonitoring supplemented with individualized, culturally tailored telephone-based nurse case management will have greater effects on blood pressure reduction and stroke recurrence and, while it will be more costly, it will also be more cost-effective than home blood pressure telemonitoring alone. Results of this study will provide strong empirical evidence to inform clinical guidelines and practice, which may lead to reductions in stroke disparities in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Black or Hispanic
* Age 18 years or older
* English or Spanish speaking
* Patients who have had an ischemic or hemorrhagic stroke
* Modified Rankin scale score of ≤ 3
* Average screening SBP ≥ 140 mm Hg from three BP readings taken at two separate visits with a validated automated device
* Receiving care at the study site for at least 6 months and planning to continue receiving care at the site for the next two years.

Exclusion Criteria:

* Being deemed unable to comply with the study protocol (either self-selected or by indicating during screening that he/she could not complete all requested tasks including using the HBPTM or interacting with the NCM if he/she were to be randomized to the intervention group)
* Participation in other clinical trials
* Diagnosis of cognitive dysfunction or significant psychiatric comorbidity (as indicated in medical record)
* Patients with upper arm circumference ≥ 52 cm, the maximum limit of the extra-large BP cuff
* Diagnosis of dialysis or end stage renal disease
* Relocating out of area or extended travel during study period
* Significant verbal speech impairment; unable to participate in intervention telephone sessions
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2014-04-18 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
12-month systolic blood pressure (SBP) change | Baseline, 12 months

SECONDARY OUTCOMES:
24-month stroke recurrence | 24 months
Cost-effectiveness for reducing SBP at 12 months | 12 months
Cost-effectiveness for reducing stroke recurrence at 24 months | 24 Months

OTHER OUTCOMES:
Change in other stroke risk factors | 6, 12, 24 months
  lipids, blood glucose
Change in health behaviors | 6, 12, 24 months
  diet, physical activity, medication adherence, weight loss
Antihypertensive medication intensification | 6, 12, 24 months
  adding, changing dose, or changing class of medications

CONTACTS AND LOCATIONS:
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Ogedegbe G, Teresi JA, Williams SK, Ogunlade A, Izeogu C, Eimicke JP, Kong J, Silver SA, Williams O, Valsamis H, Law S, Levine SR, Waddy SP, Spruill TM. Home Blood Pressure Telemonitoring and Nurse Case Management in Black and Hispanic Patients With Stroke: A Randomized Clinical Trial. JAMA. 2024 Jul 2;332(1):41-50. doi: 10.1001/jama.2024.6609. PMID 38842799
- [Derived] Spruill TM, Williams O, Teresi JA, Lehrer S, Pezzin L, Waddy SP, Lazar RM, Williams SK, Jean-Louis G, Ravenell J, Penesetti S, Favate A, Flores J, Henry KA, Kleiman A, Levine SR, Sinert R, Smith TY, Stern M, Valsamis H, Ogedegbe G. Comparative effectiveness of home blood pressure telemonitoring (HBPTM) plus nurse case management versus HBPTM alone among Black and Hispanic stroke survivors: study protocol for a randomized controlled trial. Trials. 2015 Mar 15;16:97. doi: 10.1186/s13063-015-0605-5. PMID 25873044